CLINICAL TRIAL: NCT03112863
Title: Comparison of the Cosmetic Effects of Bakuchiol and Retinol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1015536
Record Dates: First submitted 2017-03-27; First posted 2017-04-13 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Wrinkle; Photoaging
MeSH Terms: interventions — bakuchiol; Vitamin A

STUDY DESIGN:
Intervention Model Description: Double blind randomized study comparing the effect of bakuchiol and retinoid
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bakuchiol (Experimental): Bakuchiol 0.5% applied to face twice daily
  Interventions: Drug: Bakuchiol
- Retinol (Active Comparator): 0.5% retinol applied to face nightly
  Interventions: Drug: Retinol

INTERVENTIONS:
Drug: Bakuchiol — This group will receive bakuchiol
  Other Names: Bakuchiol 0.5%
  Arms: Bakuchiol
Drug: Retinol — This group will receive retinol
  Other Names: Retinol %
  Arms: Retinol

SUMMARY:
Subjects will be assigned to a retinoid cream or bakuchiol to compare the cosmetic effects. This will take place over a 12 week period.

DETAILED DESCRIPTION:
Bakuchiol is a phytochemical that has demonstrated cutaneous antiageing effects when applied topically. Early studies have suggested that bakuchiol is a functional analogue of topical retinoids, as both compounds have been shown to induce similar gene expression in the skin and lead to improvement of cutaneous photodamage. No in vivo studies have compared the two compounds for efficacy and side-effects.

The aim of this study is to compare the cosmetic effects of Bakuchiol to Retinol over a 12-week period.

ELIGIBILITY:
Inclusion Criteria:

• Individuals aged 30-55

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant or breast feeding women
* Prisoners
* Those with acne, eczema, seborrheic dermatitis, rosacea or polycystic ovarian syndrome
* Those who have used isotretinoin in the last 6 months
* Those who have used products containing salicylic acid, beta hydroxyl acids or vitamins A, C, or E in the last 14 days
* Those who have used topical antibiotics or topical retinoids in the last 30 days
* Those who are currently smoking or have smoked within the past 3 years.
* Those who have had a recent surgical or cosmetic procedure in the last 3 months that can affect facial wrinkles or facial hyperpigmentation, such as botulinum toxin injections, chemical peels, laser based therapies to the face, or face lift surgeries

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Department of Dermatology, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bakuchiol | Retinol
Started | 21 | 23
Completed | 21 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Bakuchiol 21 participants were analyzed Retinol 23 participants were analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Bakuchiol | Retinol | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — We did not include ethnicity data in this study.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 21 | 23 | 44
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Wrinkle Appearance
Description: Assessed using image analysis based assessment of wrinkle severity (depth and length).
  The primary outcome measure was image-analysis-based assessment of wrinkle severity and pigmentation at 12 weeks.
Time Frame: 12 week
Population: 21 participants were analyzed in the Bakuchiol group and 23 participants were analyzed in the Retinol group.
Measure: Number; unit: percentage of reduced fine wrinkles
Arm/Group | Bakuchiol | Retinol
Number analyzed (Participants) | 21 | 23
percentage of reduced fine wrinkles | 19.0 | 23.2

2. Primary Outcome: Percentage of Participants With Change in Appearance of Skin Pigmentation
Description: Assessed using image analysis based assessment of facial pigment
Time Frame: 12 week
Population: Pigmentation was assessed through clinical grading and through facial analysis of the surface area of involvement and overall pigment intensity.
Measure: Number; unit: percentage of participants
Arm/Group | Bakuchiol | Retinol
Number analyzed (Participants) | 21 | 23
percentage of participants | 59 | 44

3. Secondary Outcome: Number of Reports of Stinging, Burning, Itching
Description: Subjective tolerability assessment of stinging, burning, itching. Secondary outcome measures included redness, participant-reported tolerability (itching, burning and stinging) and in-person clinical assessments (pigmentation, scaling and erythema) throughout the study.
Time Frame: Assessed at Week 4, 8, and 12.
Measure: Number; unit: reports
Arm/Group | Bakuchiol | Retinol
Number analyzed (Participants) | 21 | 23
reports | 0 | 0

4. Secondary Outcome: Number of Reports of Facial Erythema Assessment
Description: Image analysis based assessment of facial erythema
Time Frame: week 4, week 8 and week 12
Measure: Number; unit: reports
Arm/Group | Bakuchiol | Retinol
Number analyzed (Participants) | 21 | 23
reports | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Subjects were no assessed for SAE or Mortality.
Arm/Group | Bakuchiol | Retinol
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/21 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT03112863/Prot_000.pdf
  • Informed Consent Form (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT03112863/ICF_001.pdf